CLINICAL TRIAL: NCT00451256
Title: Clinical Study to Assess the Safety and Efficacy of ex-Vivo Vein Graft Exposure to AVI-5126 in Coronary Artery By-Pass Grafting to Reduce Clinical Graft Failure
Brief Title: Safety and Efficacy Study of AVI-5126 When Used on Vein Grafts Before Use in Heart by-Pass Graft Surgery (CABG)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol-defined outcome in terms of efficacy would not be achieved.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AVI-5126-25
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Cardiovascular Disease; Coronary Artery Bypass
Keywords: coronary artery bypass; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AVI-5126

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AVI-5126

SUMMARY:
For some people who have heart by-pass surgery, the vein that is used to by-pass a blockage will, after some time, become narrowed and possibly blocked. AVI-5126 blocks a gene that is believed to be responsible for the events in the blood vessel that cause this narrowing. Therefore, exposing the vein to AVI-5126 before it is attached to the coronary artery may result in less problems with these vein grafts later on. This study will determine if this procedure is both safe and effective.

DETAILED DESCRIPTION:
Coronary artery bypass (CABG) is a common procedure employed for life-threatening cardiovascular disease. While bypass surgery is effective in restoring blood flow in the short-term, 30 to 50 percent of venous bypass grafts eventually become blocked or fail. Within the first year after a CABG procedure, it is estimated that between 15 and 30% of saphenous vein grafts fail (i.e., ≥ 75% reduction in flow within the graft), due to intimal hyperplasia at the anastomosis sites. There is currently no approved treatment to prevent venous graft failure. These patients may frequently undergo a second bypass surgery if the extent of graft failure(s) is sufficiently severe to lead to uncontrolled angina pectoris. It is clear that a second CABG procedure in a patient represents a higher operative mortality rate than the first procedure. Venous graft failure in CABG is a major unmet medical-surgical problem.

AVI has previously focused some of its Neugene® products in the area of preventing cardiovascular stenosis. This application of antisense targeted to to inhibit the c-myc gene has previously been demonstrated to prevent sequelae of intimal hyperplasia following endovascular injury. The purpose of this study is to evaluate whether immersion of the excised saphenous vein in a novel anti-c-myc antisense drug (AVI-5126) solution will prevent subsequent graft failure at 1 year, compared to physiological saline (placebo) prior to graft anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is a suitable candidate for aortocoronary bypass (CABG) procedure. Subjects undergoing CABG procedure without the use of coronary artery bypass (off pump) are preferred. However, subjects requiring coronary artery bypass will not be excluded from the study
* Female subjects of childbearing potential must have a documented negative serum pregnancy test within 2 days before the CABG procedure
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits
* Subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Subject will have valve replacement or repair during CABG procedure
* Subject has a poor quality donor vessel (poor or turbulent flow, varicose)
* Subject has a known left ventricular ejection fraction of <35%
* Subject has had a percutaneous coronary intervention (PCI) for coronary artery disease treatment 30 days prior to CABG
* Subject has a PCI planned during the 30 days immediately following the CABG procedure
* Subject has chronic atrial fibrillation
* Subject has a known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, or sensitivity to contrast media which cannot be adequately pre-medicated
* Subject has chronic renal insufficiency (i.e., serum creatinine >180 mmol/L) or co-morbid illness which precludes follow-up angiography
* Subject has history of a stroke or transient ischemic attack within the prior 6 months
* Subject has an active peptic ulcer or has had clinically significant upper or lower GI bleeding within the prior 6 months
* Subject has a history of a bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has a non-cardiac illness imposing substantial operative mortality
* Subject has a concurrent medical condition resulting in a life expectancy of less than 3 years
* Subject is currently participating in an investigational drug or another device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety of 10µM AVI-5126 immersion of excised saphenous vein segments prior to CABG compared to immersion in the Placebo at Day 14 and Months 1, 3, 6, 9, and 12 after CABG.

SECONDARY OUTCOMES:
to evaluate if immersion of excised saphenous vein in 10µM AVI-5126 prior to CABG reduces graft failure when compared to immersion in Placebo 12 months after CABG

CONTACTS AND LOCATIONS:
Locations (1):
- Kiev, Ukraine